CLINICAL TRIAL: NCT05082168
Title: Capnodynamic Monitoring of Cardiorespiratory Function in Patients Admitted to the Intensive Care Unit With COVID-19 Infection, Sepsis and Following Cardiac Surgery
Brief Title: Capnodynamic Monitoring of Cardiorespiratory Function in Critically Ill Patients
Acronym: PROFICIENT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South West Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Anders Aneman, Conj Professor UNSW, Director ICU Research, Senior Staff Specialist, South West Sydney Local Health District
Other Study IDs: 2020/ETH00778
Record Dates: First submitted 2021-09-20; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Acute Respiratory Infection; Sepsis; Postoperative Respiratory Distress
MeSH Terms: conditions — Sepsis | interventions — Echocardiography; Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Respiratory tract infection: Patients diagnosed with viral or bacterial pneumonia and admitted to ICU for mechanical ventilatory support
  Interventions: Device: Capnodynamic monitoring
- Sepsis: Patients diagnosed with sepsis and admitted to ICU for mechanical ventilatory support
  Interventions: Device: Capnodynamic monitoring
- Cardiac surgery: Patients admitted to ICU for mechanical ventilatory support following cardiac surgery
  Interventions: Device: Capnodynamic monitoring

INTERVENTIONS:
Device: Capnodynamic monitoring — In patients fully synchronized with mechanical ventilation, the capnodynamic method calculates the effective pulmonary blood flow, the end-expiratory lung volume and estimates the mixed venous oxygen saturation. The capnodynamic method uses short inspiratory or expiratory pauses to induce small changes in CO2 concentration the enable the mole balance to be resolved for the capnodynamic equation:
  ELV x [(FACO2(n)-FACO2(n-1)] = delta(n) x EPBF [CvCO2(n)] - VTCO2.
  Other Names: thermodilution cardiac output measurement; echocardiography; blood gas analyses

SUMMARY:
Capnodynamic monitoring has the potential to offer continuous and non-invasive measurements of heart and lung function in patients requiring ventilation in an intensive care setting. Since mechanical ventilation with full patient synchronization is commonly used in ICU, capnodynamic monitoring can be immediately embedded in clinical care and compared to current methods of monitoring cardiac output, lung volumes and oxygen delivery. This observational study will explore capnodynamic monitoring in mechanically ventilated patients with a range of cardiorespiratory compromise.

DETAILED DESCRIPTION:
This study aims to:

1. compare the estimation of cardiac output (CO) using the capnodynamic method (COEPBF) with contemporary reference methods;
2. compare the estimation of mixed venous oxygen saturation (SmvO2) with invasively obtained blood gas analyses;
3. generate observational data on end-expiratory lung volume (EELV) when ventilator settings, and in particular PEEP, are changed;
4. combine 1-3 to provide a physiological construct of cardiorespiratory function

ELIGIBILITY:
Inclusion Criteria:

Respiratory tract infection:

1. confirmed or highly suspected viral or bacterial pneumonia
2. meeting ARF or ARDS criteria as outlines in the most recent Berlin ARDS consensus statement
3. age 18 years or above
4. arterial and central venous catheters have been inserted or will be inserted as part of routine clinical management
5. mechanical ventilation via an endotracheal tube is expected to continue for the day beyond day of admission
6. adequate transthoracic echocardiographic winds are available to measure the velocity time integral in the left ventricular outflow tract
7. analgosedation is administered as part of routine management of residual neuromuscular blockaded initiated outside ICU OR the administration of analgosedation and/or neuromuscular blockers at doses that achieve full patient-ventilator synchrony are considered part of routine clinical management

Sepsis:

1. admitted to ICU with a provisional or established diagnosis of septic shock as defined by the Sepsis-3 criteria
2. age 18 years or above
3. arterial and central venous catheters have been inserted or will be inserted as part of routine clinical management
4. mechanical ventilation via an endotracheal tube is expected to continue for at least another two hours
5. adequate transthoracic echocardiographic winds are available to measure the velocity time integral in the left ventricular outflow tract
6. analgosedation is administered as part of routine management of residual neuromuscular blockaded initiated outside ICU OR the administration of analgosedation and/or neuromuscular blockers at doses that achieve full patient-ventilator synchrony are considered part of routine clinical management
7. the administration of a fluid bolus (250 ml or 500 ml) is indicated as judged by the medical officer supervising routine management

Cardiac surgery:

1. admitted to ICU following cardiac surgery using cardiopulmonary bypass
2. age 18 years and above
3. arterial, central venous and pulmonary arterial catheters have been inserted or will be inserted as part of routine clinical management
4. mechanical ventilation via an endotracheal tube is expected to continue for at least another two hours
5. analgosedation is administered as part of routine management of residual neuromuscular blockade initiated intraoperatively OR the administration of analgosedation and/or neuromuscular blockers at doses that achieve full patient-ventilator synchrony are considered part of routine clinical management
6. the administration of a fluid bolus (250 ml or 500 ml) is indicated as judged by the medical officer supervising routine postoperative management

Exclusion Criteria:

In all cohorts:

1. age under 18 years
2. known pregnancy
3. arterial and central venous catheters are not indicated as part of routine care
4. known severe valvulopathy
5. ongoing or imminent need for mechanical circulatory support
6. severe haemodynamic instability with imminent transfer for intervention(s) outside ICU
7. patient is not for full active management in ICU
8. patient is not expected to live beyond the day of admission
9. patient is re-admitted to ICU within the same index hospital admission
10. it is not possible to achieve full patient-ventilator synchrony

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU for mechanical ventilation with a diagnosis of viral/bacterial pneumonia, sepsis or following cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between capnodynamic effective pulmonary blood flow and cardiac output measured by pulmonary artery thermodilution or echocardiography | Through study completion, an average of 1 year
  Capnodynamic measurements of effective pulmonary blood flow are compared with contemporaneously obtained cardiac output measurements using clinical reference methods
Correlation between capnodynamic estimates of mixed venous oxygen saturation and blood gas analysis of blood obtained from the pulmonary artery pulmonary. | Through study completion, an average of 1 year
  Capnodynamic estimates of mixed venous oxygen saturation are compared with contemporaneously obtained blood gases from the pulmonary artery catheter
Prediction by capnodynamic monitoring of combined changes in end expiratory lung volume and effective pulmonary blood flow to assess changes in pulmonary gas exchange during various levels of PEEP | Through study completion, an average of 1 year
  At three different levels of PEEP, the interactions between end expiratory lung volume and effective pulmonary blood flow will be assessed and correlated to changes in arterial partial pressure of oxygen and carbon dioxide

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit, Liverpool Hospital, South Western Sydney Local Health District, Liverpool, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request, IPD may be shared if fully compliant with HREC requirements and European GRDP regulations

REFERENCES:
- [Derived] Keleher E, Iftikhar H, Schulz LF, McCanny P, Austin D, Stewart A, O'Regan W, Hallback M, Wallin M, Aneman A. Capnodynamic monitoring of lung volume and pulmonary blood flow during alveolar recruitment: a prospective observational study in postoperative cardiac patients. J Clin Monit Comput. 2023 Dec;37(6):1463-1472. doi: 10.1007/s10877-023-01033-1. Epub 2023 May 27. PMID 37243954
- [Derived] Schulz L, Stewart A, O'Regan W, McCanny P, Austin D, Hallback M, Wallin M, Aneman A. Capnodynamic monitoring of lung volume and blood flow in response to increased positive end-expiratory pressure in moderate to severe COVID-19 pneumonia: an observational study. Crit Care. 2022 Jul 31;26(1):232. doi: 10.1186/s13054-022-04110-0. PMID 35909174